CLINICAL TRIAL: NCT06537973
Title: The Effect of Individualized Care and Counseling Given to Primiparous Mothers in the Postpartum Period on Maternal Attachment, Maternal Self-Efficacy and Maternal Function: Randomized Controlled Trial
Brief Title: This Study Aimed to Examine the Effects of Individualized Care and Counseling Given to Mothers in the First Trimester of Pregnancy on Maternal Attachment, Maternal Self-efficacy and Maternal Function.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Nergis KARAMAN, Principal Investigator, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Necmettin EU-42
Record Dates: First submitted 2024-07-29; First posted 2024-08-05 (Actual); Last update posted 2024-08-05 (Actual); Status verified 2024-07

CONDITIONS: Maternal Behavior; Self Efficacy; Maternal Care Patterns

STUDY DESIGN:
Intervention Model Description: Parallel group (experiment-control) randomized controlled experimental
Masking Description: Since the researcher must provide training and manage the process, researcher and participant blinding cannot be done.
  Blinding in data entry; Randomization will be done by an independent researcher outside the scope of the research and the list created will be hidden from the researcher and the participants. Participants will not be informed about which group they are in until the intervention begins.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): In the first 48 hours after birth; A single-session training including postpartum care, breastfeeding and baby care will be given to mothers in the hospital room where they are hospitalized, practices will be taught and mothers will be encouraged to perform the practices.
  2nd week; Counseling will be provided to mothers who have previously been trained by contacting them via phone call.
  4th week; Phone calls will be planned with mothers, ABBÖ will be implemented, and the counseling and support provided will continue.
  6th week; A telephone interview will be planned with the mothers, MBÖ, EÖÖÖ and BAFÖ will be applied, an evaluation will be made and consultancy will be provided on the issues they need.
  8th week; A phone call will be planned with the mothers, an evaluation will be made, care plans will be maintained and counseling will be provided.
  12th week; Mothers will be contacted via phone and the MBÖ, EÖYÖ and BAFÖ scales will be applied as a posttest.
  Interventions: Other: İndividualized care education
- Control Group (No Intervention): The researchers will not provide any training or counseling to the mothers other than the standard care and services offered in the hospital. In order to ensure equality, a prepared training booklet will be given to mothers in the control group.

INTERVENTIONS:
Other: İndividualized care education — A single session of training will be given to the mothers in the experimental group. In addition, the mother will be provided with counseling by the researcher at any time she wishes. The aim is to increase the mother-infant bonding levels and self-efficacy of the mothers, who will be supported by the care plans that will be created based on Swanson's Theory of Care, and to adapt more easily to the role of motherhood, by evaluating them with the help of check-lists after the observations.
  Arms: Experimental group

SUMMARY:
Purpose of the research:

This study aimed to examine the effects of individualized care and counseling given to mothers in the first trimester after birth on maternal attachment, maternal self-efficacy and maternal function.

In this context, the hypotheses of the research are as follows:

1. Individualized care and counseling does not have a significant effect on the level of maternal attachment.
2. Individualized care and counseling does not have a positive effect on mothers' self-efficacy perceptions.
3. Individualized care and counseling does not have a significant effect on the gain of maternal function.

The study consists of experimental and control groups. The mothers of the experimental group will be interviewed in the 2nd, 4th, 6th, 8th and 12th postpartum weeks, and various surveys will be administered through counseling.

Control group mothers will not be given any training or counseling by the researcher other than the standard care and services offered in the hospital. The measurement tools applied to the experimental group mothers will be simultaneously applied to the control group mothers.

DETAILED DESCRIPTION:
Data Collection Tools: In this study, Introductory Information Form, Mother-Infant Attachment Scale, Maternal Attachment Scale (MAS), Parent Self-Efficacy Scale (PSS) and Barkin Maternal Functioning Scale (MFFS) were used as data collection tools.

Introductory Information Form: It is a form consisting of a total of 12 questions, prepared by the researcher as a result of literature review, to be applied to pregnant women and evaluating the socio-demographic (7 questions) and obstetric characteristics (5 questions) of pregnant women.

Mother-to-Infant Bonding Scale (Mother-to-Infant Bonding Scale): The scale, which allows the mother to express the feelings she feels towards her baby with a single word, was developed by Taylor et al. in 2005. The original name of the scale is Mother-Infant Attachment Scale. The scale was adapted into Turkish by Karakulak Aydemir in 2009. Mother-Baby Attachment Scale is a 4-point Likert type scale consisting of 8 items. According to the results of the guidance, the items Loving, Neutral/feeling nothing, Joyful, Dislike and Protective are placed under the first factor, and the items Angry, Disappointment and Anger are placed under the second factor. Responses consisting of four options are scored between 0-3. The lowest score that can be obtained from the scale is 0, while the highest score is 24. The responses to the items in the scale are as follows; 0 = A lot, 1 = A lot, 2 = A little, 3 = Not at all. In the evaluation, items 1, 4 and 6 express positive emotional expressions, while items 2, 3, 5 and 7 express negative emotional expressions and are scored reversely. An increase in the score obtained from the scale indicates a mother-infant attachment problem.

Maternal Attachment Scale (MBS): The scale measuring maternal feelings and behaviors that show love was developed by Muller in 1994. The scale was first applied to mothers at 30-40 days postpartum, and then in the fourth and eighth months. The scale, adapted to Turkish society as a result of the study of Kavlak and Şirin in 2009, was tested on mothers with one- and four-month-old babies. The expressions of the one-dimensional scale, consisting of a total of 26 items in the four-point likert type, were determined as always=a (4 points), often=b (3 points), sometimes=c (2 points) and never=d (1 point).The lowest score to be obtained from the scale is 26 and the highest score is 104. A high score indicates high maternal attachment. Muller found the Cronbach Alpha coefficient of the scale to be 0.85, 0.76 and 0.85, respectively, and Şirin and Kavlak found it to be 0.77 in mothers with one-month-old babies and 0.82 in mothers with four-month-old babies.

Parental Self-Efficacy Scale (EÖS): The scale was developed by Kılıçaslan in 2007 to determine the personal judgments of parents of their first babies aged 3-6 months regarding their competence in the parental role.It is a 5-point likert-type scale consisting of 18 items. The scale has 5 sub-dimensions. Items 11, 12, 13, 16, 18 indicate baby's needs, items 1, 5, 6, 9 indicate parenting skills, items 2, 4, 10, 17 indicate baby's mental state, items 7, 8, 15 indicate baby's disorders, and items 3 and 14 indicate baby's emotions. The responses to the items in the scale are listed as strongly agree, agree, undecided, disagree and strongly disagree. The scale is scored on a scale from 1 to 5. In case of opposite statements, the scores will be reversed and the calculation will be made. The Cronbach Alpha value of the scale was found to be 0.852.

Barkin Maternal Function Scale (BAFÖ): The Turkish validity and reliability of the scale developed by Barkin in 2009 to evaluate the functional status of the mother after birth was conducted by Aydın in2016. The seven-point likert type scale consists of a total of 16 questions. The responses on the scale are numbered between 0 and 6. 0 means strongly disagree, 1 means disagree, 2 means slightly disagree, 3 means undecided, 4 means slightly agree, 5 means agree, 6 means strongly agree.The lowest score that can be obtained from the scale is 0 and the highest score is 96. Evaluation is made based on the total score. A high score means that the maternal function is high. The Barkin Maternal Function Scale, which is recommended to be used starting from 6-10 weeks postpartum and up to two years, includes five subscales: self-care, maternal psychology, baby care, social support and adaptation to motherhood. Barkin found the Cronbach Alpha value of the scale to be 0.87, and Aydın found it to be 0.73.

ELIGIBILITY:
Inclusion Criteria:

* Being primiparous
* Having a vaginal birth
* Having given birth at term
* Being 18 years or older
* Having a single, healthy baby
* Must be at least a primary school graduate
* The mother does not have a diagnosed chronic or psychiatric disease.
* Volunteering to participate in the study

Exclusion Criteria:

* • Having a history of risky pregnancy

  * Participated in any birth preparation training program
  * The mother shows signs of mental or physical illness (self-report/clinical diagnosis).
  * Inability to communicate effectively with the mother
  * The baby has a health problem

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 54 (Estimated)
Dates: Start 2024-07-31 (Estimated); Primary Completion 2024-08-05 (Estimated); Study Completion 2024-09-15 (Estimated)

PRIMARY OUTCOMES:
Mother-to-Infant Bonding Scale (ABBÖ) | It will be applied in the 4th and 12th weeks.
  It is a scale that allows the mother to express the feelings she feels towards her baby with a single word. It is a 4-point Likert type scale consisting of 8 items. Responses consisting of four options are scored between 0-3. The lowest score that can be obtained from the scale is 0, while the highest score is 24.
Maternal Attachment Scale (MBS) | It will be applied in the 6th and 12th weeks.
  It is a one-dimensional scale consisting of a total of 26 items in a four-point Likert type that measures maternal feelings and behaviors that show love. The expressions were determined as "always (a) (4 points)", "often (b) (3 points)", "sometimes (c) (2 points)" and "never (d) (1 point)". The lowest score to be obtained from the scale is 26 and the highest score is 104. A high score indicates high maternal attachment.
Parental Self-Efficacy Scale (EÖSÖ) | It will be applied in the 6th and 12th weeks.
  It is an 18-item, 5-point Likert type scale developed to determine parents' personal judgments about their competence in the parental role. The answers to the items on the scale are listed as "Totally Agree", "Agree", "Undecided", "Disagree" and "Strongly Disagree".
Barkin Maternal Function Scale (BAFÖ) | It will be applied in the 6th and 12th weeks.
  The seven-point Likert type scale, developed to evaluate the functional status of the mother after birth, consists of a total of 16 questions. Responses on the scale are expressed as 0 "strongly disagree", 1 "disagree", 2 "somewhat disagree", 3 "undecided", 4 "somewhat agree", 5 "agree", 6 "completely agree". The lowest score that can be obtained from the scale is 0 and the highest score is 96. Evaluation is made based on the total score. A high score means that the maternal function is high.

SECONDARY OUTCOMES:
Maternal Attachment Scale (MBS) | It will be applied in the postpartum weeks.
  It is a one-dimensional scale consisting of a total of 26 items in a four-point Likert type that measures maternal feelings and behaviors that show love. The expressions were determined as "always (a) (4 points)", "often (b) (3 points)", "sometimes (c) (2 points)" and "never (d) (1 point)". The lowest score to be obtained from the scale is 26 and the highest score is 104. A high score indicates high maternal attachment.
Parental Self-Efficacy Scale (EÖSÖ) | It will be applied in the 12th week.
  It is an 18-item, 5-point Likert type scale developed to determine parents' personal judgments about their competence in the parental role. The answers to the items on the scale are listed as "Totally Agree", "Agree", "Undecided", "Disagree" and "Strongly Disagree".
Barkin Maternal Function Scale (BAFÖ) | It will be applied in the 6th week.
  The seven-point Likert type scale, developed to evaluate the functional status of the mother after birth, consists of a total of 16 questions. Responses on the scale are expressed as 0 "strongly disagree", 1 "disagree", 2 "somewhat disagree", 3 "undecided", 4 "somewhat agree", 5 "agree", 6 "completely agree". The lowest score that can be obtained from the scale is 0 and the highest score is 96. Evaluation is made based on the total score. A high score means that the maternal function is high.

CONTACTS AND LOCATIONS:
Overall Officials: Emel EGE Prof. Dr., Study Director — Necmettin Erbakan University
Locations (1):
- Necmettin Erbakan University, Konya, Meram, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
After the study is completed, the parts to be shared will be discussed again and a decision will be made.